CLINICAL TRIAL: NCT05721924
Title: Comparing The Effectiveness Of Pericapsular Nerve Group (PENG) Block Versus Supra-Inguinal Fascia Iliaca Compartment Block(S-FICB) In Reducing Positional Pain During Neuraxial Anaesthesia In Hip Fractures Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FF-2022-336
Record Dates: First submitted 2023-01-26; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Hip Fractures
Keywords: Hip Fractures Patients Going For Internal Fixation
MeSH Terms: conditions — Hip Fractures | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: The recruited patients will be randomly divided into two groups via stratified randomization based on patient's hips fractures classification. Intra-articular fractures involving fractures within the hip joint. While extra-articular fractures are those fractures outside the capsule of the hip joint which are intertrochanteric and subtrochanteric. Two envelopes will be prepared which is intra-articular and extra-articular fractures envelope. In each envelope, there will be 10 "A" blocks and 10 "B" blocks.
Who Masked: Participant, Care Provider
Masking Description: The recruited patients and the attending anaesthetist will be blinded to the type of block provided for the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pericapsular nerve group (PENG) block (Active Comparator): The pericapsular nerve group (PENG) block is an ultrasound-guided approach, first described by Giron-Arango et al. for the blockade of the articular branches of the femoral, obturator and accessory obturator nerves that provide sensory innervation to the anterior hip capsule.
  Interventions: Procedure: Pericapsular nerve group (PENG) block
- Supra-inguinal fascia iliaca compartment (S-FICB) block (Active Comparator): A supra-inguinal fascia iliaca compartment block (S-FICB), a 3 in 1 block involving femoral nerve , lateral femoral cutaneous nerve and obturator nerve.
  Interventions: Procedure: Supra-inguinal fascia iliaca compartment (S-FICB) block

INTERVENTIONS:
Procedure: Pericapsular nerve group (PENG) block — In PENG group, the patient will be given PENG block 30mls of 0.2% ropivacaine
  Arms: Pericapsular nerve group (PENG) block
Procedure: Supra-inguinal fascia iliaca compartment (S-FICB) block — Patients in group B (S-FICB group) will be supra-inguinal fascia iliaca compartment block 30mls of 0.2% ropivacaine
  Arms: Supra-inguinal fascia iliaca compartment (S-FICB) block

SUMMARY:
Fractures in and around the hip are common in the elderly and most of them required early surgical fixation. Hip fractures are accompanied with a considerable amount of pain. Based on National Orthopaedic Registry Malaysia (NORM), spinal/neuraxial anaesthesia makes up 66.3%, is the preferred mode of anaesthesia. Severe pain associated with fractured hip often results in difficulty during positioning for neuraxial anaesthesia and hence it is extremely challenging to position the patients in sitting or lateral position for neuraxial anaesthesia procedures. A supra-inguinal fascia iliaca compartment block (S-FICB), a 3 in 1 block involving femoral nerve , lateral femoral cutaneous nerve and obturator nerve. It is famous technique among anaesthesiologist to treat immediate and postoperative pain in hip fractures patients. The pericapsular nerve group (PENG) block is an ultrasound-guided approach, first described by Giron-Arango et al. in 2018 for the blockade of the articular branches of the femoral, obturator and accessory obturator nerves that provide sensory innervation to the anterior hip capsule. It is an alternative regional anaesthesia technique for the management of acute pain after hip fracture. The goal of this clinical trial is to compare the effectiveness of (PENG) block vs (S-FICB) block in reducing positional pain during neuraxial block in patients going for elective internal fixation of neck of femur fractures. And investigators's hypothesis is PENG block is as effective as S-FICB in reducing positional pain during neuraxial block in patients going for elective internal fixation of neck of femur fractures.

DETAILED DESCRIPTION:
The recruited participants will be randomly divided into two groups via stratified randomization based on participants's neck of femur fractures classification. Intra-articular fractures involving fractures within the hip joint. While extra-articular fractures are those fractures outside the capsule of the hip joint which are intertrochanteric and subtrochanteric. Two envelopes will be prepared which is intra-articular and extra-articular fractures envelope. In each envelope, there will be 10 "A" blocks and 10 "B" blocks. Researcher will draw from the particular envelope and thus Group A will be receiving PENG Block 30mls of 0.2% ropivacaine; Group B where the S-FICB will be given 30mls of 0.2% ropivacaine which will be prepared by researcher.

The demographic data of the participants which include age, gender, height, weight, body mass index (BMI), ASA status, diagnosis and type of surgery will be recorded in the data collection sheet. Standard monitoring devices will be applied to all paricipants such as automatic non-invasive blood pressure (NIBP), electrocardiograph (ECG), and pulse oximetry (SPO2) will be recorded at baseline. Baseline pain scores (PS0) at rest and on movement (15° passive elevation) as PS0m will be recorded in the data collection sheet before PENG block or S-FICB administration and recorded on numeric pain rating scale (NRS). Pain score will be assessed via numerical pain rating scale (NRS) which the scale is composed of 0 (no pain at all) to 10 (worst imaginable pain). The pain score will be categorised into mild pain (score of 1-4); moderate pain (score of 5-7) and severe pain (score of 8-10). The block will be performed by a single operator who has been trained to perform the block by a certified trained regional anaesthesia specialist (credentialed by performing at least 20 successful PENG and S-FICB block). The operator will undergo a probationary phase under supervision of a regional anaesthetist in UKMMC by performing at least 5 PENG and 5 S-FICB in HUKM. A report will be written to the committee regarding capability and safety of the operator before starting the study.

In the PENG group, the participant will be placed in supine position and the monitoring devices will be applied as mentioned earlier and the baseline parameters will be recorded. The block will be administered under ultrasound guidance with a curvilinear probe/linear probe locating the iliopubic eminence, iliopsoas tendon and femoral artery. Stimuplex® needle, an echogenic needle that enables use of nerve stimulation and visualized under ultrasound in performing peripheral nerve blocks 100 mm 22 G will be advanced from lateral to medial approach until the needle tip reach the plane between the iliopsoas tendon and periosteum which is between anterior inferior iliac spine and iliopubic eminence. Next, 30 mls of local LA agent ropivacaine 0.2% will be injected. There will be total of 60 mg of Ropivacaine (maximum dose 3mg/kg). The 30 mls of LA solution (ropivacaine 0.2%) will be injected in 5 mls increments while observing for adequate fluid spread under ultrasound guided. Negative aspiration will be performed at the start of the injection and after each 5 mls of the injectate. The spread of LA below iliopsoas tendon and floating up iliopsoas tendon indicate correct LA distribution.

Participants in group B (S-FICB group) will be positioned supine with extended hip, and any abdominal pannus will be retracted by an assistant or heavy tape. The anterior superior iliac spine (ASIS) will be located and the ultrasound probe will be placed slightly inferior and medial to ASIS with a parasagittal orientation and more perpendicular to the inguinal ligament. The iliacus muscle will be identified superficial to the ilium and the hyperechoic fascia iliaca will be identified on the superficial border of the muscle. Superficial to the fascia iliaca, there will be abdominal wall muscles meet those of the lower extremity at the inguinal ligament. The Stimuplex® needle will be inserted from the caudal directed cephalad in in-plane approach until the needle tip reach the fascia iliaca plane. Then, 1-2 mls of saline or local anaesthetic will be injected to confirm spread between the hyperechoic fascia iliaca and the more heterogeneous iliacus muscle beneath it. The 30 mls of LA solution (ropivacaine 0.2%) will be injected in 5 mls increments while observing for adequate fluid spread under ultrasound guided. Negative aspiration will be performed at the start of the injection and after each 5 mls of the injectate.

In both the groups, the vital signs of participants, NIBP and ECG, respiratory rate (RR) and SpO2 will be evaluated at 5 minute intervals for 30 minute after the injection. Pain score will be assessed at 30 minute post bock during rest (PSPB) and on movement at 15° passive elevation (PSPBm). Pain score will be assessed via numerical pain rating scale (NRS) as explained above. If any patient has NRS> 4/10 then will be considered as failed block and will be dropped out from the study. The failed block participants will be managed by the attending anaesthetists in charged based on the standard protocol and rescue analgesia with IV fentanyl 50mcg will be given to the participant. All participants will be carefully observed to detect any symptoms of LA toxicity such as peri-oral and tongue numbness, dizziness, tinnitus, visual disturbances, seizure, unconscious, respiratory depression and cardiovascular depression as per standard protocol. Any paricipant who developed LA toxicity will be treated based on the standard management and will be dropped out from the study.

After 30 minutes of observation following the block for both the groups, the participants will be pushed into the dedicated operating room and the spinal anaesthesia (SA) or combined spinal epidural anaesthesia (CSE) will be performed by the attending anaesthetists in charge based on the standard protocol. The attending anaesthetist will be blinded to the type of block provided for the participants.

During the positioning for neuraxial anaesthesia, the pain score during the positioning will be assessed via NRS and the ease of positioning will be graded by the attending anaesthetist with the scale of 0-3 (0 = unable to position, 1= participant has abnormal posturing due to pain and require support for positioning, 2= mild discomfort but does not require support for positioning, 3=optimal condition where the participant is able to position himself/ herself without pain) as adopted from Jadon A. et al. Subsequent management of the participants throughout the surgery will be carried out by the attending anaesthetists as per standard protocol throughout the perioperative period. Post neuraxial anaesthesia the paricipants will be rated for satisfaction score via Likert scale for the block been given.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II and III
* Hip fractures such as neck of femur (not older than 2 weeks and have persistent pain)

Exclusion Criteria:

* Patients contraindicated to peripheral nerve blocks
* Patients with history of chronic pain
* Patients with significant cognitive impairment
* Patients with known allergic to study medications

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain score | 30 minutes after intervention
  Baseline pain scores (PS0) at rest and on movement (15° passive elevation) as PS0m will be recorded in the data collection sheet before PENG block or S-FICB administration and recorded on numeric pain rating scale (NRS).Pain score will be assessed via numerical pain rating scale (NRS) which the scale is composed of 0 (no pain at all; the best scoring) to 10 (worst imaginable pain; the worst scoring). The pain score will be categorised into mild pain (score of 1-4); moderate pain (score of 5-7) and severe pain (score of 8-10). Pain score will be assessed at 30 minute post bock during rest (PSPB) and on movement at 15° passive elevation (PSPBm). Pain score during positioning during neuraxial anaesthesia also will be recorded.

SECONDARY OUTCOMES:
Ease of positioning during neuraxial anaesthesia | 30 minutes after intervention
  The ease of positioning will be graded by the attending anaesthetist with the scale of 0-3 (0 = unable to position, 1= patient has abnormal posturing due to pain and require support for positioning, 2= mild discomfort but does not require support for positioning, 3=optimal condition where the patient is able to position himself/ herself without pain)(The highest the score; the better the positional scoring)
Patient satisfaction toward the block being given | 30 minutes after neuraxial anaesthesia being given
  Post neuraxial anaesthesia the patients will be rated for satisfaction score via Likert scale for the block been given.(The higher the score; the better satisfaction toward the intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Canselor Tuanku Muhriz, Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur, Malaysia